CLINICAL TRIAL: NCT02166424
Title: The Synchronized Trial on Expectant Mothers With Depressive Symptoms by Omega-3 PUFAs (SYNCHRO)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tokyo Medical University (Other)
Collaborators: China Medical University, Taiwan (Other); Japan Society for the Promotion of Science (JSPS) (Unknown); University of Toyama (Other); Chiba University (Other); National Center for Child Health and Development (Unknown)
Responsible Party: Principal Investigator, Daisuke Nishi, Assistant Professor, Tokyo Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SYNCHRO-RCT
Record Dates: First submitted 2014-06-15; First posted 2014-06-18 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Pregnancy; Depression
Keywords: Pregnancy; Depression; omega-3 fatty acids
MeSH Terms: conditions — Depression | interventions — Docosahexaenoic Acids; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 polyunsaturated fatty acids (Active Comparator): 1200mg eicosapentaenoic acid (EPA) and 600mg docosahexaenoic acid (DHA) daily
  Interventions: Dietary Supplement: Omega-3 polyunsaturated fatty acids
- olive oil (Placebo Comparator): 2880mg olive oil daily
  Interventions: Dietary Supplement: Olive oil

INTERVENTIONS:
Dietary Supplement: Omega-3 polyunsaturated fatty acids
  Other Names: 1200mg EPA and 600mg DHA daily
  Arms: Omega-3 polyunsaturated fatty acids
Dietary Supplement: Olive oil
  Other Names: 2880mg olive oil daily
  Arms: olive oil

SUMMARY:
The present study aims to examine the efficacy and safety of omega-3 polyunsaturated fatty acids for pregnant women with depressive symptoms.

DETAILED DESCRIPTION:
Maternal depression can have a significant harmful influence on both mothers and children. Considering the possibility of adverse effects of antidepressants and previous meta-analyses showing the positive effects of omega-3 polyunsaturated fatty acids (PUFAs) supplementation in reducing depressive symptoms, omega-3 PUFAs may provide a safe strategy. The investigators evaluate efficacy and safety of omega-3 PUFAs for pregnant women with depressive symptoms. (Participants who skipped taking supplements for more than 7 days will be excluded from a per protocol analysis.)

ELIGIBILITY:
Inclusion Criteria:

1. pregnant women aged 20 years or older
2. between 12-24 weeks gestation
3. a Japanese conversational ability in Japan site or a Mandarin conversational ability in Taiwan site to understand the scope of the present trial and to provide written consent for study participation
4. planned to take assessments after childbirth
5. an Edinburgh Postnatal Depression Scale (EPDS) score is 9 or more
6. to have good physical health judged by obstetricians.

Exclusion Criteria:

1. history and current suspicion of psychosis or bipolar I disorder or substance-related disorder or eating disorder or personality disorder
2. Serious psychiatric symptoms such as self-harm behavior or in need of rapid psychiatric treatment
3. difficult to expect a normal birth (ex: fetal malformation etc.)
4. having a history of bleeding disorder such as von Willebrand's Disease
5. regular treatment with aspirin or warfarin within the last 3 months
6. a smoking habit of ≥40 cigarettes per day
7. regular treatment with ethyl icosapentate or regular consumption of omega-3 PUFA supplements within the last 3 months
8. a habit of eating fish as a main dish ≥4 times per week.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
total score of the Hamilton Rating Scale for Depression (HAMD) | Twelve weeks

SECONDARY OUTCOMES:
total score of HAMD | 4-6 weeks after childbirth
major depressive disorder (MDD) as determined by the depression module of the Mini International Neuropsychiatric Interview (MINI) | Twelve weeks, 4-6 weeks after childbirth
total scores on the Edinburgh Postnatal Depression Scale (EPDS) | Twelve weeks, 4-6 weeks after childbirth
total score of the Beck Depression Inventory Ⅱ(BDI-Ⅱ) | Twelve weeks, 4-6 weeks after childbirth
omega-3 fatty acids concentrations in erythrocytes | Tweve weeks, 4-6 weeks after childbirth
brain-derived neurotrophic factor (BDNF) in serum | Twelve weeks, 4-6 weeks after childbirth
estrogen in plasma | twelve weeks, 4-6 weeks after childbirth
oxytocin in plasma | twelve weeks, 4-6 weeks after childbirth
progesterone in plasma | twelve weeks, 4-6 weeks after childbirth
human chorionic gonadotropin (hCG) in plasma | twelve weeks, 4-6 weeks after childbirth
phospholipase A2 in plasma | twelve weeks, 4-6 weeks after childbirth

OTHER OUTCOMES:
gestational age | at childbirth
gestational diabetes mellitus | 4-6 weeks after childbirth
gestational hypertension or preeclampsia | 4-6 weeks after childbirth
induced labour | at childbirth
estimated blood loss | at childbirth
cesarean section | at childbirth
operative vaginal delivery | at childbirth
birthweight | at childbirth
one minute apger | 4-6 weeks after childbirth
5-minute apgar | 4-6 weeks after childbirth
neonatal intensive care unit admission | 4-6 weeks after childbirth
cholesterol | twelve weeks and 4-6 weeks after childbirth

CONTACTS AND LOCATIONS:
Overall Officials: Daisuke Nishi, M.D., Ph.D., Principal Investigator — Tokyo Medical University; Kuan-Pin Su, M.D., Ph.D., Principal Investigator — China Medical Univeristy
Locations (4):
- Japan (3):
  - Toda Chuo Women's Hospital, Toda, Saitama
  - National Center for Child Health and Development, Setagaya City, Tokyo
  - Tokyo Medical University, Shinjyuku-ku, Tokyo
- China Medical University, Taichung, Taiwan

REFERENCES:
- [Derived] Nishi D, Su KP, Usuda K, Chiang YJ, Guu TW, Hamazaki K, Nakaya N, Sone T, Sano Y, Tachibana Y, Ito H, Isaka K, Hashimoto K, Hamazaki T, Matsuoka YJ. The synchronized trial on expectant mothers with depressive symptoms by omega-3 PUFAs (SYNCHRO): Study protocol for a randomized controlled trial. BMC Psychiatry. 2016 Sep 15;16(1):321. doi: 10.1186/s12888-016-1031-2. PMID 27630014